CLINICAL TRIAL: NCT06450106
Title: A Phase 1 Dose Escalation Study of STM-416p Administered Intraoperatively to Patients Undergoing Radical Prostatectomy
Brief Title: Study of STM-416p Administered to Patients Undergoing Radical Prostatectomy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SURGE Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STM-416p-201
Record Dates: First submitted 2024-06-02; First posted 2024-06-10 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Intraoperative; Dose escalation; Open-label; STM-416; Resiquimod; Toll-like receptor 7/8; Radical prostatectomy; Robotic prostatectomy; Immunotherapy; STM-416p; PSA; R848; Hydrogel
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- STM-416p (Experimental): STM-416p
  Interventions: Drug: STM-416p

INTERVENTIONS:
Drug: STM-416p — STM-416p monotherapy

SUMMARY:
A Study of STM-416p Administered Intraoperatively to Patients Undergoing Radical Prostatectomy

DETAILED DESCRIPTION:
A Phase 1 Dose Escalation Study of STM-416p Administered Intraoperatively to Patients Undergoing Radical Prostatectomy

ELIGIBILITY:
Inclusion Criteria:

1. Males aged 18 years or older at time of informed consent.
2. Have a histologically confirmed diagnosis of prostate cancer, and are scheduled to undergo radical prostatectomy within 28 days of screening.
3. Grade Group 2-5.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2 at Screening.
5. Have adequate organ and bone marrow function at screening.
6. Able to understand and be willing to sign an Institutional Review Board/Ethics Committee-approved written informed consent document

Exclusion Criteria:

1. Have an invasive malignancy, other than the disease under study.
2. Anticipated to require the use of a drain after radical prostatectomy.
3. Received any other anticancer therapy (e.g., including but not limited to chemotherapy, biologic therapy, immunotherapy, targeted therapy, endocrine therapy, radiation therapy, intravesical therapy ) within 28 days.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition as those used in the STM-416p formulation including poloxamer 407 and sodium hyaluronate.
5. History of allogeneic organ transplant.
6. History of primary immunodeficiency.
7. QTc interval >470 msec at Screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) [Safety and Tolerability] | 21 Days
  Incidence of dose-limiting toxicities (DLTs) over the first 21-days of study treatment
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Time on trial up to 90 days
  Incidence of serious adverse events (SAEs), and adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

SECONDARY OUTCOMES:
Pharmacokinetics of STM-416p | Day 0, post 24 hours, post 48 hour
  Maximum plasma concentration (Cmax) of resiquimod (R848) in patient blood
Pharmacodynamics of STM-416p in blood circulating cytokines | Day 0, post 24 hours, post 48 hours, post 21 days
  Pharmacodynamic assessments in plasma and urine will be listed and summarized by dose level
Assess surgical wound healing | Day 7, Day 21
  Assessment of wound healing scored according to a modified ASEPSIS method

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Arizona Urology Specialists, Tucson, Arizona
  - University of Florida, Gainesville, Florida
- Australia (2):
  - Australian Prostate Center, Melbourne N., Victoria
  - Epworth HealthCare, Melbourne N., Victoria

IPD SHARING:
Plan to Share IPD: No